CLINICAL TRIAL: NCT01969253
Title: A Prospective Observational Study of Lymphedema in Breast Cancer With Axillary Lymph Node Dissection (ALND)
Brief Title: A Prospective Observational Study of Lymphedema in Breast Cancer With Axillary Lymph Node Dissection
Status: Completed | Type: Observational
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, So-Youn Jung, Medical Doctor, National Cancer Center, Korea
Other Study IDs: NCC-1210181-2
Record Dates: First submitted 2013-08-14; First posted 2013-10-25 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer, Axillary Lymph Node Dissection, Lymphedema
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Over the past few years, several studies have been made on various outcomes about the incidence of lymphedema. Because the outcomes can be came out differently each study by measurement, criteria, treatment period, treatment method and morbid extremities of lymphedema. Therefore it is required for understanding about the incidence, risk factor and physical progress for to be treated and prevented of lymphedema. Also it is necessary that to understand characteristics of lymphedema measurements and to establish diagnostic criteria of lymphedema through comparative study.

The aim of this study was to analyze the incidence and risk factor of lymphedema through prospectively observation, and to determine effects on the quality of life of lymphedema after breast cancer surgery with ALND.

DETAILED DESCRIPTION:
Primary Objectives:

- To analyze incidence rate of lymphedema using tape measurements, perometre, bioimpedance, spectroscopy.

Secondary Objectives:

* To determine the risk factor of lymphedema in postoperative breast cancer.
* To understand that lymphedema has an effect on quality of life and physical function in postoperative breast cancer.
* To complete uestionnaire about physical and quality of life in postoperative breast cancer with ALND patients.

ELIGIBILITY:
Inclusion Criteria:

* Older than 20 years old
* Patient who underwent unilateral Breast Cancer surgery with ALND
* Informed consent must to be signed

Exclusion Criteria:

* Previous history of breast cancer
* History of abnormality or vascular disease in upper extremity
* Patients with other serious systemic illness (renal failure, hepatic dysfunction, congestive heart failure, neurological or psychological impairment) that would confound the study or impair the patients' ability to participate.
* History of infection on upper extremity
* History of corticosteroid use on whole body for any reason
* Inability to provide informed consent (e.g. dementia or severe cognitive impairment)

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective study is observational study that focused on incidence of lymphedema in breast cancer patients. Annually six hundred patients have received treatment of breast cancer from the breast cancer center at National Cancer Center in Korea. Among of them, two hundred patients have received surgical treatment with axillary dissection. About four hundred patients were recruited consecutively for enrollment from May 2012 to December 2013.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2012-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the incidence of lymphedema in upper arm after ALND | Up to 1year
  In this study, we evaluated the incidence of lymphedema in upper arm using tape measurement, perometre and bioimpedance spectroscopy during pre,post-operative visit, 3, 6, 9month and 1year clinical follow-up.

SECONDARY OUTCOMES:
To Evaluate quality of life using questionnaire | Up to 1year
  * European Organization for Research and Treatment of Cancer(EORTC) the 30-item version of the core Quality of Life Questionnaire (EORTC QLQ C30)
  * EORTC Quality of Life Questionnaire - Breast Cancer Module (EORTC QLQ BR23)
Physical assess | Up to 1year
  * Questionnaire: Disabilities of the arm shoulder and hand using (DASH)
  * Physical examination

CONTACTS AND LOCATIONS:
Overall Officials: So-Youn Jung, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea